CLINICAL TRIAL: NCT00424372
Title: A LONG-TERM STUDY TO EVALUATE SAFETY AND EFFICACY STUDY OF PREGABALIN IN THE TREATMENT OF POSTHERPETIC NEURALGIA.
Brief Title: A Long-Term Study To Evaluate Safety And Efficacy Of Pregabalin For Postherpetic Neuralgia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: A0081121
Record Dates: First submitted 2007-01-18; First posted 2007-01-19 (Estimated); Results first posted 2009-09-28 (Estimated); Last update posted 2021-08-27 (Actual); Status verified 2021-07

CONDITIONS: Neuralgia, Postherpetic
MeSH Terms: conditions — Neuralgia, Postherpetic | interventions — Pregabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- pregabalin (Experimental)
  Interventions: Drug: pregabalin

INTERVENTIONS:
Drug: pregabalin — Dosage: 150-600 mg/day (75-300 mg bid), oral administration, Treatment duration: 52 weeks

SUMMARY:
To evaluate the safety of the long-term use of pregabalin.

ELIGIBILITY:
Inclusion Criteria:

* Patients who completed the 13-week treatment of postherpetic neuralgia in Study A0081120.
* Patients must be able to understand and cooperate with study procedures and have signed a written informed consent prior to entering the study.

Exclusion Criteria:

* Patients who experienced serious adverse events in the preceding study (A0081120) that were determined by the investigator or the study sponsor to be causally related to the study medication.
* Patients exhibiting treatment non-compliance in the preceding study (A0081120)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2007-01-12 (Actual); Primary Completion 2008-08-19 (Actual); Study Completion 2008-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (33):
- Japan (33):
  - National Hospital Organization Nagoya Medical Center, Nagoya, Aichi-ken
  - Kobayashi Clinic, Urayasu, Chiba
  - Okabe Hospital, Kasuya-gun, Fukuoka
  - Gunma Pain Clinic Hospital, Maebashi, Gunma
  - Takasaki Pain Clinic, Takasaki, Gunma
  - Asahikawa Pain Clinic Hospital, Asahikawa, Hokkaido
  - Kamui Pain Clinic, Asahikawa, Hokkaido
  - Sapporo Asabu Clinic, Sapporo, Hokkaido
  - Higashi Sapporo Hospital, Sapporo, Hokkaido
  - Seimei Clinic, Akashi, Hyōgo
  - Uchida Pain Relief Clinic, Amagasaki, Hyōgo
  - National Hospital Organization Himeji Medical Center, Himeji, Hyōgo
  - National Hospital Organization Kobe Medical Center, Kobe, Hyōgo
  - Nakamura Clinic, Kobe, Hyōgo
  - National Hospital Organization Sagamihara National Hospital, Sagamihara, Kanagawa
  - Suzuki Pain Clinic, Yokohama, Kanagawa
  - Hajiri Pain Clinic, Yokohama, Kanagawa
  - National Hospital Organization Yokohama Medical Center, Yokohama, Kanagawa
  - Sendai Pain Clinic, Sendai, Miyagi
  - Nakamura Hospital, Beppu, Ohita
  - Kawaguchi Kogyo General Hospital, Kawaguchi, Saitama
  - Kinoshita Clinic, Tokorozawa, Saitama
  - Tokyo Women's Medical University Center East, Arakawa-ku, Tokyo
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - Mitaka Pain Clinic, Mitaka, Tokyo
  - Toriumi Pain Clinic, Nakano-ku, Tokyo
  - Kanto Medical NTT East Corporation, Shinagawa-ku, Tokyo
  - Naganuma Pain Clinic, Shinagawa-ku, Tokyo
  - Tokyo Women's Medical University Hospital, Shinjuku-ku, Tokyo
  - Mukai Clinic, Fukuoka
  - KM Pain Clinic, Fukuoka
  - Otsuki Sleep Clinic, Fukushima
  - Hasumi Pain Clinic, Saitama

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081121&StudyName=A%20Long-Term%20Study%20To%20Evaluate%20Safety%20And%20Efficacy%20Of%20Pregabalin%20For%20Postherpetic%20Neuralgia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 126 subjects who completed the 13-week treatment regimen in the preceding double-blind Study A0081120 and had no serious adverse events or issues with compliance were enrolled to this study.
Groups:
- Pregabalin: Subjects initiated study drug at 75 mg in the evening of Day 1, and then 75 mg BID (150 mg/day) for 1 week from Day 2. Subsequent dose modifications were based on subjects' safety and efficacy response and the maximum doses were 150 mg BID (300 mg/day) for subjects with low creatinine clearance (CLcr) (30 < CLcr ≤ 60 mL/min) and 300 mg BID (600 mg/day) for subjects with normal CLcr (CLcr > 60 mL/min).
Period: Overall Study
Arm/Group | Pregabalin
Started | 126
Completed | 95
Not Completed | 31
Not completed — Death | 1
Not completed — Adverse Event | 18
Not completed — Lack of Efficacy | 6
Not completed — Withdrawal by Subject | 4
Not completed — Protocol Violation | 1
Not completed — Health deterioration | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pregabalin
Number analyzed (Participants) | 126
Age, Customized [Number; unit: Subjects]
  >= 18 and < 45 years | 1
  >= 45 and < 65 years | 19
  >=65 years | 106
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55
  Male | 71

OUTCOME MEASURES:

1. Primary Outcome: Summary of Adverse Events
Description: Number of subjects with all causality adverse events, serious adverse events, severe adverse events, adverse events resulted in discontinuation, dose reduced or temporary discontinuation. Subjects are counted only once per treatment in each row.
Time Frame: 52 weeks
Population: Safety population: all subjects who took at least 1 dose of study medication.
Measure: Number; unit: subjects
Arm/Group | Pregabalin
Number analyzed (Participants) | 126
subjects
  Subjects with adverse events | 124
  Subjects with serious adverse events | 14
  Subjects with severe adverse events | 5
  Subjects discontinued due to adverse events | 17
  Dose reduced or temporary discontinuation | 34

2. Secondary Outcome: Short-Form McGill Pain Questionnaire the Efficacy of Change: Sensory Score
Description: Score ranges: 0-33. Higher scores indicate more severe pain. Baseline: The last evaluation on or before Day 1 of double-blind for subjects that took pregabalin in double-blind and last visit <= Day 1 of open-label for subjects that took placebo in double-blind. Endpoint: The last evaluation during dose adjustment/maintenance step of open-label.
Time Frame: 52 weeks
Population: Full Analysis Set, N = Number of subjects assessed
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Pregabalin
Number analyzed (Participants) | 126
score on scale
  Baseline | 11.3 (7.0)
  Week 52: number analyzed (Participants) | 94
  Week 52 | 5.1 (5.6)
  Endpoint | 6.7 (7.1)
  Change from Baseline to Endpoint | -4.8 (5.9)

3. Secondary Outcome: Short-Form McGill Pain Questionnaire the Efficacy of Change: Affective Score
Description: Score ranges: 0-12. Higher scores indicate more severe pain. Baseline: The last evaluation on or before Day 1 of double-blind for subjects that took pregabalin in double-blind and last visit <= Day 1 of open-label for subjects that took placebo in double-blind. Endpoint: The last evaluation during dose adjustment/maintenance step of open-label.
Time Frame: 52 weeks
Population: Full Analysis Set, N = Number of subjects assessed
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Pregabalin
Number analyzed (Participants) | 126
score on scale
  Baseline | 3.4 (3.1)
  Week 52: number analyzed (Participants) | 94
  Week 52 | 1.0 (1.8)
  Endpoint | 1.7 (2.7)
  Change from Baseline to Endpoint | -1.8 (2.8)

4. Secondary Outcome: Short-Form McGill Pain Questionnaire the Efficacy of Change: Total Score
Description: Score ranges: 0-45. Higher scores indicate more severe pain. Baseline: The last evaluation on or before Day 1 of double-blind for subjects that took pregabalin in double-blind and last visit <= Day 1 of open-label for subjects that took placebo in double-blind. Endpoint: The last evaluation during dose adjustment/maintenance step of open-label.
Time Frame: 52 weeks
Population: Full Analysis Set, N = Number of subjects assessed
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Pregabalin
Number analyzed (Participants) | 126
score on scale
  Baseline | 14.7 (9.7)
  Week 52: number analyzed (Participants) | 94
  Week 52 | 6.1 (7.2)
  Endpoint | 8.2 (9.6)
  Change from Baseline to Endpoint | -6.5 (8.4)

5. Secondary Outcome: Short-Form McGill Pain Questionnaire the Efficacy of Change: Present Pain Intensity
Description: Score ranges: 0-5. Higher scores indicate more severe pain. Baseline: The last evaluation on or before Day 1 of double-blind for subjects that took pregabalin in double-blind and last visit <= Day 1 of open-label for subjects that took placebo in double-blind. Endpoint: The last evaluation during dose adjustment/maintenance step of open-label.
Time Frame: 52 weeks
Population: Full Analysis Set, N = Number of subjects assessed
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Pregabalin
Number analyzed (Participants) | 126
score on scale
  Baseline | 2.8 (1.0)
  Week 52: number analyzed (Participants) | 94
  Week 52 | 1.4 (0.9)
  Endpoint | 1.7 (1.1)
  Change from Baseline to Endpoint | -1.1 (1.1)

6. Secondary Outcome: Short-Form McGill Pain Questionnaire the Efficacy of Change: Visual Analog Scale
Description: Ranges: 0-100 mm. Larger scale indicate more severe pain. Baseline: The last evaluation on or before Day 1 of double-blind for subjects that took pregabalin in double-blind and last visit <= Day 1 of open-label for subjects that took placebo in double-blind. Endpoint: The last evaluation during dose adjustment/maintenance step of open-label.
Time Frame: 52 weeks
Population: Full Analysis Set, N = Number of subjects assessed
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Pregabalin
Number analyzed (Participants) | 126
mm
  Baseline | 62.0 (19.0)
  Week 52: number analyzed (Participants) | 94
  Week 52 | 28.3 (22.9)
  Endpoint | 33.7 (25.6)
  Change from Baseline to Endpoint | -28.3 (23.8)

ADVERSE EVENTS:
Time Frame: 52 weeks
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Pregabalin
Serious Adverse Events (participants affected / at risk) | 15/126
Other Adverse Events (participants affected / at risk) | 98/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=126)
Atrial fibrillation (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Gastroduodenal ulcer (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Pneumonia (Infections and infestations) | 1
Heat stroke (Injury, poisoning and procedural complications) | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1
Open fracture (Injury, poisoning and procedural complications) | 1
Radius fracture (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 2
Occult blood (Investigations) | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Completed suicide (Psychiatric disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Malignant palate neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=126)
Retinal haemorrhage (Eye disorders) | 7
Visual acuity reduced (Eye disorders) | 7
Constipation (Gastrointestinal disorders) | 12
Diarrhoea (Gastrointestinal disorders) | 12
Nausea (Gastrointestinal disorders) | 7
Oedema peripheral (General disorders) | 22
Nasopharyngitis (Infections and infestations) | 34
Fall (Injury, poisoning and procedural complications) | 9
Weight increased (Investigations) | 19
Arthralgia (Musculoskeletal and connective tissue disorders) | 7
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 7
Dizziness (Nervous system disorders) | 36
Headache (Nervous system disorders) | 7
Somnolence (Nervous system disorders) | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.